CLINICAL TRIAL: NCT03754439
Title: Minimising the Adverse Physiological Effects of Transportation on the Premature Infant
Acronym: TRiPs
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Nottingham (Other)
Responsible Party: Sponsor
Other Study IDs: 18015
Record Dates: First submitted 2018-11-12; First posted 2018-11-27 (Actual); Last update posted 2018-11-27 (Actual); Status verified 2018-11

CONDITIONS: Prematurity; Transfer Injury; Brain Injuries; Intraventricular Hemorrhage; Vibration; Exposure; Noise Exposure
MeSH Terms: conditions — Premature Birth; Brain Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Inborn: * Infants born within Nottingham University hospitals
  * < 32 weeks gestational age
  * < 72 hours old
  Interventions: Behavioral: Physiological changes to noise and vibration exposure
- Transported: - Infants born outside of Nottingham University Hospitals or transferred between units Phase 1 < 32 weeks gestational age and <72 hours old Phase 2 any gestation and age
  Interventions: Behavioral: Physiological changes to noise and vibration exposure

INTERVENTIONS:
Behavioral: Physiological changes to noise and vibration exposure — Physiological parameters (HR, RR, Sats, NIRS) will be observed during a period of stay on the neonatal unit (Inborn group) or during ambulance transportation (Transported group) whilst simultaneous measurement of noise and vibration exposure. Urine will be collected during the first 24, 48 and 72 hours post exposure for biochemical markers of brain injury (S100B) and stress (Cortisol)

SUMMARY:
Centralisation of neonatal intensive care has led to an increase in postnatal inter-hospital transfers within the first 72 hours of life. Studies have shown transported preterm infants have an increased risk of intraventricular haemorrhage compared to inborns. The cause is likely multi-factorial, however, during the transportation process infants are exposed to noxious stimuli (excessive noise, vibration and temperature fluctuations), which may result in microscopic brain injury. However, there is a paucity of evidence to evaluate the effect of noise and vibration exposure during transportation.

In this study the investigators aim to quantify the level of vibration and noise as experienced by a preterm infant during inter-hospital transportation in ground ambulance in the United Kingdom

Secondary aims of the study are to:

i) measure the physiological and biochemical changes that occur as a result of ambulance transportation (ii) quantify microscopic brain injury through measurement of urinary S100B and other biomarkers (iii) evaluate the development of intraventricular haemorrhage on cranial ultrasound iv) monitor vibration and sound exposure, using a prototype measuring system, during neonatal transport using both a manikin and a small cohort of neonatal patients.

v) evaluate vibration and sound exposure levels using an updated transportation system modified to reduce effects.

DETAILED DESCRIPTION:
There were 50 000 premature births in the United Kingdom (UK) and this number is increasing each year due to changes in demographics of the childbearing population with a trend towards increasing maternal age, increased uptake in fertility treatments and a greater number of medically induced deliveries. This has resulted in a greater risk of preterm delivery. Significant advances in neonatal intensive care have led to better survival rates with more preterm infants surviving at the extremes of gestational age. However, this is not without significant co-morbidity in terms of increased incidence of respiratory disease, cerebral palsy, learning difficulties and behavioural problems in surviving infants. The long term effect of impairment in cognitive functioning has led to an increased incidence of special education needs (one to one support, special schools), lower scores of cognitive ability (e.g. reading & maths), a higher rate of school failure and lower up take of higher education in early adulthood in these infants.

Due to the increasing preterm birth rate year strategies to reduce this level of morbidity are of great importance to public health care. In 2003, neonatal services were reorganised into managed clinical network leading to the development of hospitals of different specialist levels of care working together with the aim to improve provision of quality care and neonatal outcomes. Although this change in practice has led to an increase in survival, the level of neurodisability has remained the same. Furthermore, the number of neonatal inter-hospital has subsequently increased (10,000 in 2010 to 16,000 in 2016) with the necessity to move premature infants to higher level centres for on-going care but also the need to move infants due to lack of available cots at higher level centres.

Neonatal transport has been associated with significant morbidity in terms of severe intraventricular haemorrhage (IVH). A large study of 69 000 very low birth weight infants based in the USA showed infants who undergo inter-hospital transportation within the first 72 hours of life, a period when infants are most vulnerable to IVH, are 75% more likely to develop any IVH and 44% more likely to develop severe IVH compared to inborn non-transported infants. Severe IVH has been associated with both short and long term neurological morbidity and mortality. It has been estimated 50 to 80% of survivors with severe IVH develop cerebral palsy and 70% have cognitive impairment. Mild IVH, although not significantly associated with severe impairment, has been shown result in lower developmental scores at school age, with a higher percentage of infants requiring educational support compared to infants who never developed IVH.

Given the significant lifelong impact of severe IVH on premature infants, their families and society, current practice needs to be stratified to reduce the risk associated with transportation. The causation of this additional morbidity is unknown and likely to be multifactorial. However, studies that have accounted for risk factors known to be associated with IVH, such as, low birth weight and intubation using multivariable regression models have still found an association between transport and IVH, which raises the question whether the physical process of transportation itself contributes to the development of IVH.

During transportation infants are exposed to both excessive vibration and noise. Studies have shown in healthy adults excessive vibration is associated with adverse health effects, such as, fatigue, headaches, circulatory disturbance and neurological disorders. Studies have shown neonates are exposed to vibration levels during neonatal transport to be in the range of 0.4-5.6m/s2, which would be deemed extremely uncomfortable by International Standards Organization (ISO) 2631. However, a weakness of all these studies accessing vibration levels during transport is in the location of the vibration sensor during measurement, which is either placed on the mattress or incubator and therefore may not give a true reflection of the vibration exposure the neonate's head endures.

Currently, there is a paucity of evidence to evaluate the effect of vibration on neonates especially during transportation. Cerebral blood flow can be monitored via near infra-red spectrometry (NIRS), which is a real time and non-invasive technique. Soul et al demonstrated that continuous monitoring of regional cerebral oxygenation with NIRS can be correlated with changes in systemic blood pressure and provide insight into the fluctuating nature of cerebral pressure in preterm infants and hence identify infants at risk of cerebral pathology. NIRS monitoring during ambulance transfer would allow real time assessment of the cerebral perfusion during ambulance transfer. Additionally, simultaneous vibration and noise measurement will allow correlation of exposure levels with changes in cerebral perfusion.

In addition, exposure to excessive sound, like vibration, has been shown to have adverse effects in healthy adults and neonates. Excessive noise has been shown to increase heart rate (HR), increase blood pressure, increase respiratory rates (RR) and alter sleep cycles in both term and preterm infants. Premature infants have decreased autonomic self-regulatory mechanisms and are unable to adapt to loud noxious stimuli, which predisposes them to physiological instability. This instability can potentially result in fluctuations in cerebral blood flow, which could increase the risk of bleeds.

Although a small number of studies have documented vibration (although of the incubator) and noise exposure during transportation, none of the studies have correlated the level of exposure with physiological changes or biochemical markers of neurological injury. Correlation of vibration exposure as experienced by the neonatal head and noise exposure within the incubator will allow the investigators to plan interventional strategies aimed at reducing both vibration and noise exposure. Overall, by reducing these noxious stimuli the investigators aim to reduce both subtle neurological injury and IVH to improve long term neurodevelopmental outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Infant < 32 weeks gestation (Phase 1) or any neonatal patient (Phase 2)
* Less than 72 hours of age
* With written maternal consent

Exclusion Criteria:

* Lethal and/or major congenital abnormality known at study entry
* No realistic prospect of survival
* No informed consent
* Maternal death

Max Age: 4 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Neonatal patients
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2018-10-31 (Actual); Primary Completion 2020-07-31 (Estimated); Study Completion 2020-07-31 (Estimated)

PRIMARY OUTCOMES:
Vibration | An average of 90 minutes
  Vibration exposure levels during ambulance journey or inborn measurement for period as experienced by the infant's head & incubator (m/s2)
Noise | An average of 90 minutes
  Sound exposure levels during the ambulance journey or inpatient measurement period both inside and outside the incubator (dB)

SECONDARY OUTCOMES:
Intraventricular haemorrhage | Until discharge from hospital, on average 3-4 months after admission.
  Development of intraventricular haemorrhage on cranial ultrasound scan, Scans will be taken pre and 24 hours post transfer for transported groups. Both transported and inborn infants will have their routine cranial ultrasound scan results documented on day 1, 3, 7 and d28 or discharge cranial ultrasound, whichever came first, from time of birth until discharge from hospital.
Heart rate (beats per minute) | an average of 90 min
  Heart rate will be measured either during the ambulance journey or inpatient measurement period including following journery undertaken in modified transport system
Pulse oximetery (oxygen saturation %) | An average of 90 min
  Oxygen saturations will be measured either during the ambulance journey or inpatient measurement period including following journery undertaken in modified transport system
Respiratory rate (breaths per minute) | An average of 90 min
  Respiratory rate will be measured every 15 minutes either during the ambulance journey or inpatient measurement period including following journery undertaken in modified transport system
Near infrared spectroscopy (regional oxygen saturations) | An average of 90 min
  Regional oxygen saturations via NIRS will be measured either during the ambulance journey or inpatient measurement period including following journery undertaken in modified transport system
Urine biochemical measurements | 3 days
  Urine will be collected within the first 24 hours, 48 hours and 72 hours following vibration and noise exposure in the ambulance. Inborn patients will have urine collected within the first 24, 48 and 72 hours following measurement period. Urine will be used to quantify level of S100B.

CONTACTS AND LOCATIONS:
Overall Officials: Don Sharkey, MBBS, PhD, Principal Investigator — University of Nottingham
Locations (1):
- University Hospitals Nottingham NHS Trust, Nottingham, Nottinghamshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Blaxter L, Yeo M, McNally D, Crowe J, Henry C, Hill S, Mansfield N, Leslie A, Sharkey D. Neonatal head and torso vibration exposure during inter-hospital transfer. Proc Inst Mech Eng H. 2017 Feb;231(2):99-113. doi: 10.1177/0954411916680235. Epub 2017 Jan 5. PMID 28056712